CLINICAL TRIAL: NCT02711579
Title: Impact of Selective Cyclooxygenase-2 Inhibitor, Celecoxib on Cortical Excitability and Electrophysiological Property in Brain of Healthy Volunteer: Randomized, Double-blind, Placebo-controlled Study
Brief Title: Impact of Celecoxib on Electrophysiological Property in Brain of Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-1509-130-708
Record Dates: First submitted 2016-03-08; First posted 2016-03-17 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2016-12

CONDITIONS: Electrophysiologic Property of Brain
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Celecoxib for electroencephalography (Experimental): Electroencephalography will be performed before and after celecoxib administration
  Interventions: Drug: Celecoxib
- Placebo for electroencephalography (Placebo Comparator): Electroencephalography will be performed before and after placebo administration
  Interventions: Drug: Placebo
- Celecoxib for motor evoked potential (Experimental): Motor evoked potential will be measured before and after celecoxib administration
  Interventions: Drug: Celecoxib
- Placebo for motor evoked potential (Placebo Comparator): Motor evoked potential will be measured before and after placebo administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib
  Arms: Celecoxib for electroencephalography; Celecoxib for motor evoked potential
Drug: Placebo
  Arms: Placebo for electroencephalography; Placebo for motor evoked potential

SUMMARY:
the purposes of this study are to evaluate the acute electrophysiological response in brain cortex to single oral dose of celecoxib (400mg once) in healthy volunteer and the electrophysiological alteration in brain cortex by long-term treatment of celecoxib (200mg twice-daily for 7 days) in healthy volunteer

DETAILED DESCRIPTION:
Inflammatory response is considered as defense mechanism against physical or infectious insults and also prevails within the central nervous system. Following certain kinds of brain injuries (i.e trauma, ischemia, hypoxia and seizure), innate immunity and subsequent adaptive immunity subserve the robust inflammatory cascades, leading to excitatory synaptic networks. Cellular elements, such as neuron, microglia as well as inflammatory molecules (cyclooxygenase2, interleukin-1, tumor necrosis factor-alpha, etc) play essential roles in enhancing this process.

In line with these, compelling evidences in animal studies in epilepsy field indicate that celecoxib (COX-2 inhibitor) has anticonvulsant actions, although its mechanisms are not fully understood. Thus, oral administration of Celecoxib in human has a high potential to suppress the neuronal excitability. As a milestone for the big picture, current study is going to prove the changes of cortical excitability evoked by transmagnetic stimulation (TMS) and electroencephalographic properties revealed by EEG in healthy volunteer, given that power spectral analysis of EEG and several parameters of TMS , can detect the small changes of neuronal activities by celecoxib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged between 20 and 50 years.
* Signed voluntary written informed consent.
* Body mass index between 16.0 and 30.0 kg/m2.

Exclusion Criteria:

* History of cardiovascular disease (i.e. Heart disease, Stroke), hepatic disease, inflammatory bowel disease, gastrointestinal hemorrhage, or seizure(s).
* History of hypersensitivity to any medication(s) (i.e. urticaria, angioedema, shock)
* History of any kind of medication(s) within 1 week before screening.
* Presence of clinically significant electrocardiogram abnormality at screening.
* aspartate transaminase or alanine transaminase : greater than 2.0 × upper normal limit.
* Serum creatinine levels : greater than 1.5 × upper normal limit.
* Platelet counts lower than 100,000 / μL
* Serum potassium : greater than 5.5 mmol/L
* Female who is pregnant, breastfeeding, or intends to become pregnant.
* History of noncompliance with medications.
* History of alcohol abuse.
* Participation in drug study within 30 days before screening.
* Galactose intolerance

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Power spectral change by single oral dose of celecoxib (400mg once) in healthy volunteer | 4 hours after medical treatment
  Power spectrum will be measured by electroencephalography
Cortical excitability alteration in brain cortex by long-term treatment of celecoxib (200mg twice-daily for 7 days) in healthy volunteer | 7 days after medical treatment
  Cortical excitability will be measured by transmagnetic stimulation

SECONDARY OUTCOMES:
Power spectral change by celecoxib in different locations and different frequency band. | 4 hours and 7 days after medical treatment
  Power spectrum will be measured by electroencephalography

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Il Park, MD., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea